CLINICAL TRIAL: NCT05081791
Title: Effects of Exercise Therapy on Functional Capacity, Muscle Strength and Patient-reported Outcomes in Patients with Muscle Dystrophies
Brief Title: Exercise Therapy for Patients with Muscle Dystrophies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Raquel Sebio, Lecturer, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCLINIC - MD - 2021
Record Dates: First submitted 2021-09-22; First posted 2021-10-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Muscular Dystrophies
Keywords: exercise therapy; muscle strength; exercise tolerance; muscular dystrophies
MeSH Terms: conditions — Muscular Dystrophies | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Post-training assessments will be conducted by a blinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Training (Experimental): This group will engage in a 12-week exercise training program
  Interventions: Behavioral: Exercise Training
- Control group (No Intervention): Usual care. Patients in this group will be offered the same program at the end of the study

INTERVENTIONS:
Behavioral: Exercise Training — 12-week exercise training program including a combination of endurance and resistance training for 45 minutes, twice a week.
  Arms: Exercise Training

SUMMARY:
Muscular Dystrophies (MD) are a heterogeneous group of diseases characterised by muscle wasting that lead to progressive loss of function. Although exercise training has been traditionally neglected to these patients due to concerns regarding muscle damage, research has shown that exercise therapy is safe and tolerable in this population and can lead to potential gains in endurance and muscle strength, as well as other patient-reported outcomes such as health-related quality of life.Therefore, in this study, the investigators aim to examine the feasibility, tolerability and safety as well as the effects of a 12-week, exercise-training program in patients with MD on functional capacity, muscle strength, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or Genetically diagnosis of Muscular Dystrophy including Limb-Girdle type I and type II, Myotonic Dystrophy type I and type II and facioscapulohumeral dystrophy.
* Age > 18 years old
* Ability to walk independently for 10 or more metres

Exclusion Criteria:

* Inability to understand or read Spanish/Catalan.
* Patients engaging in a similar exercise-based program in the past 12 months
* Patients with severe cognitive, neurological or musculoskeletal impairment unable to participate in the exercise program
* Unstable respiratory, cardiovascular or metabolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | 1 week post-intervention
  Time consumed by the patient to raise from a chair, walk 3 meters, turn 180º, walk 3 metres back and sit down on the chair

SECONDARY OUTCOMES:
Short Physical Performance Battery | 1 week post-intervention
  Score in this test is derived from three assessments: balance, gait speed and lower limb muscle performance
Upper Body Muscle Strength | 1 week post-intervention
  Muscle strength of the biceps brachii will be assessed with a hand-held dynamometer
Lower Body Muscle Strength | 1 week post-intervention
  Muscle strength of the quadriceps will be assessed with a hand-held dynamometer
Handgrip Strength | 1 week post-intervention
  Handgrip strength will be assessed with a hydraulic dynamometer.
Health-Related Quality of Life | 1 week post-intervention
  HRQoL will be measured with the Short-Form Health Survey (SF-12). The score of the scale goes from 0 - 100, with higher scores representing better health-related quality of life.
Body Weight | 1 week post-intervention
  Body weight (kg)
Body Mass Index | 1 week post-intervention
  Body weight and height will be combined to report the results on body mass index (kg/m2)
Percentage of fat-free mass | 1 week post-intervention
  Percentage of fat-free mass will be obtained through bio-impedance analysis
Percentage of fat mass | 1 week post-intervention
  Percentage of fat mass will be obtained through bio-impedance analysis
Fatigue | 1 week post-intervention
  Fatigue will be quantified with the Brief Fatigue Inventory. The scale has 9 items with a maximal score of 10 points. Higher scores represent heavier fatigue.
Respiratory Muscle Strength | 1 week post-intervention
  Maximal Inspiratory and Expiratory Muscle Strength will be measured according to international guidelines (ATS/ERS) with a MicroRPM.
Physical Activity Levels | 1 week post-intervention
  Accelerometry-assessment of physical activity will be measured in terms of steps per day and minutes spent in light, moderate and vigorous physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain